CLINICAL TRIAL: NCT05343676
Title: Different Sonographic Modalities in Compared With PET-CT in Evaluation of Pediatric Lymphoma
Brief Title: Different Sonographic Modalities and PET-CT in Pediatric Lymphoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hager Mohammed Abdelhafiez, principle investigator, Assiut University
Other Study IDs: imaging in pediatric lymphoma
Record Dates: First submitted 2022-02-11; First posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Pediatric Lymphoma
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ultrasonography — * For assessment of LNS ( cervical , axillary and inguinal LNS ), The choice of transducer is an important consideration when evaluating lymph nodes as higher frequencies provide better resolution for superficial structures
  * For color Doppler assessment of the lymph nodes, scanning will be done using the slow frame rate, low pulse repetition frequency
  * Assessment features including lymph node location, size, shape, border, echogenicity, calcifications, necrosis or cystic change, and adjacent soft tissue edema

SUMMARY:
* To evaluate the accuracy of different sonographic modalities vs PET/CT in assessment of response to therapy in lymphoma patients: both early and late therapeutic response assessment.
* To evaluate whether imaging features of pathologic lymph nodes on PET/CT and ultrasonography have a predictive role before, during and after treatment in comparison to clinical outcome.

DETAILED DESCRIPTION:
Lymphomas are common malignancies in children [1]. Lymphomas account for about 5% to 6% of all malignancies [2] and include a number of different pathologic subtypes, which arise from the constituent cells of the immune system or from their precursor, lymphoma is now highly treatable. Imaging plays a major role in diagnosis, staging and response making surgical staging unnecessary in most cases [3].

The treatment regimen and the prognosis depend on the morphological type of lymphoma and the disease stage [4].

PET/CT using (18F) FDG is considered one of the functional imaging techniques used to assess the glucose metabolism in vivo; its use has been widely increased in evaluation of oncology patients being highly sensitive in assessment of malignancy as PET/CT can detect malignancy prior to morphological change[5].

Imaging by PET is vastly improved by combining it with CT technology. FDG-PET and CT provide functional and anatomic information, respectively. Integration of both modalities can compensate for the disadvantages of each, and the combination method outperforms , thus PET CT has a proved role for Lymphoma in adult [6].

F-FDG PET/CT is now considered the most accurate imaging modality in the management of adult lymphomas. Its value has been well documented for initial staging, at mid chemotherapy, after the end of therapy, and for assessing tumor recurrence in the follow-up [7,8].

Diagnostic information obtained from 18F-FDG PET scans changed management in 24% of pediatric oncology patients, including those with lymphoma [9].

The sensitivities of FDG-PET for the detection of nodal and extra nodal lesions of lymphoma are 92-100 and 74-78% [10].

The formation of multiple lymph node lesions in distant sites is one of the characteristics differentiating this disease from lymph node metastasis of common cancer, and thus the fact that FDG-PET allows whole-body scanning is a strong point in its favor.[11].

Ultrasonography is an imaging modality that is favored worldwide because of its precision, portability, practicality, and cost. The use of this technology to distinguish metastatic from benign cervical lymph nodes, this determination has implications for diagnosis, staging, and determining optimal treatment regimens [12].

Lymph node enlargement is a common feature of various benign and malignant disorders. It is well recognised that ultrasound is superior to palpation in detecting and characterising subcutaneous lymph nodes, various sonographic modalities can be used for lymph node evaluation, including gray-scale, color Doppler [13].

Nodal sonographic features can offer a clue for whether a lymph node contains cancer. Ultrasound provides detailed information about the internal and external features of a lymph node and demonstrates superior sensitivity and specificity in detecting malignant nodes compared with physical examination [14].

With the use of color Doppler sonography, the vasculature of the lymph nodes can also be evaluated which provides additional information about the nodes. It has become an effective way to obtain more information about the examined lymph nodes with no appreciable increase in the duration or invasiveness of the examination [15].

ELIGIBILITY:
Inclusion Criteria:

Age: 16 yrs or younger . Proved lymphoma with histopathology

Exclusion Criteria:

Hypersensitivity to 18fluorine FDG Patients

Ages: 1 Year to 16 Years | Sex: All
Age Groups: Child
Study Population: Male or female patients. Age: 16 yrs. or younger . Proved lymphoma with histopathology
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Different Sonographic Modalities in Compared with PET-CT in Evaluation of Pediatric Lymphoma | baseline
  To evaluate the accuracy of different sonographic modalities vs PET/CT in assessment of response to therapy in lymphoma patients

CONTACTS AND LOCATIONS:
Overall Officials: haisam ahmed samy, professor, Study Director — Assiut University; mohamed moamen elbaroudy, doctor, Study Director — Assiut University

REFERENCES:
- [Background] McCarten KM, Nadel HR, Shulkin BL, Cho SY. Imaging for diagnosis, staging and response assessment of Hodgkin lymphoma and non-Hodgkin lymphoma. Pediatr Radiol. 2019 Oct;49(11):1545-1564. doi: 10.1007/s00247-019-04529-8. Epub 2019 Oct 16. PMID 31620854
- [Background] Gupta A, Rahman K, Shahid M, Kumar A, Qaseem SM, Hassan SA, Siddiqui FA. Sonographic assessment of cervical lymphadenopathy: role of high-resolution and color Doppler imaging. Head Neck. 2011 Mar;33(3):297-302. doi: 10.1002/hed.21448. PMID 20652889
- [Background] Giacomini CP, Jeffrey RB, Shin LK. Ultrasonographic evaluation of malignant and normal cervical lymph nodes. Semin Ultrasound CT MR. 2013 Jun;34(3):236-47. doi: 10.1053/j.sult.2013.04.003. PMID 23768890
- [Background] Elshikh M, Moawad AW, Salem U, Klimkowski SP, Hassan T, Rao Korivi B, Jensen CT, Javadi S, Elsayes KM. Oncologic Imaging of the Lymphatic System: Current Perspective with Multi-Modality Imaging and New Horizon. Cancers (Basel). 2021 Sep 10;13(18):4554. doi: 10.3390/cancers13184554. PMID 34572781
- [Background] Kleis M, Daldrup-Link H, Matthay K, Goldsby R, Lu Y, Schuster T, Schreck C, Chu PW, Hawkins RA, Franc BL. Diagnostic value of PET/CT for the staging and restaging of pediatric tumors. Eur J Nucl Med Mol Imaging. 2009 Jan;36(1):23-36. doi: 10.1007/s00259-008-0911-1. Epub 2008 Aug 22. PMID 18719909
- [Background] Kostakoglu L, Leonard JP, Kuji I, Coleman M, Vallabhajosula S, Goldsmith SJ. Comparison of fluorine-18 fluorodeoxyglucose positron emission tomography and Ga-67 scintigraphy in evaluation of lymphoma. Cancer. 2002 Feb 15;94(4):879-88. PMID 11920454
- [Background] Jerusalem G, Beguin Y, Fassotte MF, Belhocine T, Hustinx R, Rigo P, Fillet G. Early detection of relapse by whole-body positron emission tomography in the follow-up of patients with Hodgkin's disease. Ann Oncol. 2003 Jan;14(1):123-30. doi: 10.1093/annonc/mdg011. PMID 12488304
- [Background] Wegner EA, Barrington SF, Kingston JE, Robinson RO, Ferner RE, Taj M, Smith MA, O'Doherty MJ. The impact of PET scanning on management of paediatric oncology patients. Eur J Nucl Med Mol Imaging. 2005 Jan;32(1):23-30. doi: 10.1007/s00259-004-1645-3. Epub 2004 Jul 31. PMID 15290124
- [Background] Yamamoto F, Tsukamoto E, Nakada K, Takei T, Zhao S, Asaka M, Tamaki N. 18F-FDG PET is superior to 67Ga SPECT in the staging of non-Hodgkin's lymphoma. Ann Nucl Med. 2004 Sep;18(6):519-26. doi: 10.1007/BF02984570. PMID 15515753
- [Background] Johnson SA, Kumar A, Matasar MJ, Schoder H, Rademaker J. Imaging for Staging and Response Assessment in Lymphoma. Radiology. 2015 Aug;276(2):323-38. doi: 10.1148/radiol.2015142088. PMID 26203705
- [Background] Chang DB, Yuan A, Yu CJ, Luh KT, Kuo SH, Yang PC. Differentiation of benign and malignant cervical lymph nodes with color Doppler sonography. AJR Am J Roentgenol. 1994 Apr;162(4):965-8. doi: 10.2214/ajr.162.4.8141027.
- [Background] Barrington SF, Mikhaeel NG, Kostakoglu L, Meignan M, Hutchings M, Mueller SP, Schwartz LH, Zucca E, Fisher RI, Trotman J, Hoekstra OS, Hicks RJ, O'Doherty MJ, Hustinx R, Biggi A, Cheson BD. Role of imaging in the staging and response assessment of lymphoma: consensus of the International Conference on Malignant Lymphomas Imaging Working Group. J Clin Oncol. 2014 Sep 20;32(27):3048-58. doi: 10.1200/JCO.2013.53.5229. PMID 25113771
- See also: Baba, S., Abe, K., Isoda, T. et al. Impact of FDG-PET/CT in the management of lymphoma. Ann Nucl Med 25, 701-716 (2011) — https://doi.org/10.1007/s12149-011-0549-0